CLINICAL TRIAL: NCT06692543
Title: Immunometabolic and Neuromuscular Markers of Vitality Capacity : SENIOR Protocol
Brief Title: Sedentary or Exercised : Neuromuscular and Immunometabolic Observations and Retrospection
Acronym: SENIOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: LAMHESS (Unknown); Institut de bilogie de Valrose (Unknown); INSERM-C3M (Unknown); LP2M (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 24-PP-07
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Aging
Keywords: immunity; aging; muscles; exercise; metabolism; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 2x20 people aged >55 yo, 1 group physically active, the other is physically inactive
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physically active (Experimental): Participants of this group are physically active subjects
  - V1 will take place at the Nice University Hospital, in the morning, on an empty stomach.
  After signing the consent form, the participant will have a blood sample taken (24mL), answer questionnaire and have a body assessment by bone densitometry. At the end of the appointment , the participant will wear an accelerometer and fill in his or her food intake for one week.
  - V2 (approximatly 2 weeks after V1), will take place at LAMHESS, the participant will perform neuromuscular tests on an ergometer, with high-density electromyography (HDEMG) sensors on the thighs.
  Interventions: Other: Active population
- Physically inactive (Experimental): Participants of this group are physically inactive subjects
  - V1 will take place at the Nice University Hospital, in the morning, on an empty stomach.
  After signing the consent form, the participant will have a blood sample taken (24mL), answer questionnaire and have a body assessment by bone densitometry. At the end of the appointment , the participant will wear an accelerometer and fill in his or her food intake for one week.
  - V2 (approximatly 2 weeks after V1), will take place at LAMHESS, the participant will perform neuromuscular tests on an ergometer, with high-density electromyography (HDEMG) sensors on the thighs.
  Interventions: Other: Inactive population

INTERVENTIONS:
Other: Active population — 1 blood withdraw, questionnaire and tests
  Arms: Physically active
Other: Inactive population — 1 blood withdraw, questionnaire and tests
  Arms: Physically inactive

SUMMARY:
The distinction between healthy and pathological ageing has given rise to the vitality capacity concept. Underlying the physiological aspect of ageing, vitality capacity is reflected in the neuromuscular function, metabolism, and immune and stress response. The three domains seem to deteriorate with age, except among individuals who have maintained physical activity throughout their lives. Furthermore, immune cells, particularly T lymphocytes, appear to play a key role in each dimension of vitality capacity, as well as in the mice ageing pathway. Investigators sought to determine the effect of lifelong physical activity on vitality capacity, and especially on T cell metabolism.

In this optic, fourty healthy participants over the age of 55 will be allocated to two groups: 20 who have maintained physical activity for the past 30 years, and 20 who have not. Each participant's vitality capacity will be deeply tested and compared to their physical activity background.

ELIGIBILITY:
* General Inclusion Criteria:
* Men and women > 55 years old
* Participants who are non-smokers or have been weaned for more than 3 years
* Menopausal women (confirmed for at least 6 months)
* Participants affiliated to the social security system
* Signature of informed consent
* Inclusion Criteria for the active population:
* Any person with structured aerobic physical activity (mainly involving cardiorespiratory function) on at least 3 days/week over the last 30 years without an interruption of more than 1 week in the 3 months preceding the study and without an interruption of more than 12 consecutive months over the last 30 years, as assessed by an interview conducted by an investigator specialising in physical activity;
* have a level of physical activity that meets the recommendations for physical activity in terms of the duration and intensity of weekly cardiorespiratory effort (WHO, 2020; ANSES, 2016) according to the criteria assessed by the GPAQ: at least 150 to 300 minutes per week of moderate-intensity aerobic activity (e.g., 5 days of moderate intensity activity of at least 30 minutes/day) or at least 75 to 150 minutes of sustained intensity endurance activity (e.g., 3 days of sustained activity of 25 minutes/day); or an equivalent combination of moderate and sustained intensity activities throughout the week.
* Inclusion criteria for the inactive population :
* Any person who does not meet the criteria for inclusion in the 'active' population defined above;
* Any person who has or has had a low physical intensity professional activity over the last 30 years: sedentary professional activity (work time generally spent in a seated position, such as office work) and/or a standing professional activity (work time spent standing or walking, without intense physical effort (e.g. shop assistant, hairdresser, caretaker, etc.).
* Anyone who does not practise or has not practised sport, fitness or other physical leisure activities alone or under supervision over the last 30 years, or who practises or has practised, over the last 30 years, a sport, fitness or other physical leisure activity less than or equal to 2 days a week and for a weekly period not exceeding 75 minutes.
* Anyone whose active mode of transport (cycling, walking) does not exceed an overall duration of 75 minutes per week, and whose consecutive time slots per journey are less than 10 minutes.
* Non-inclusion Criteria:
* Person suffering from a chronic illness
* Anyone who has used performance-enhancing drugs
* Anyone with a disability
* Person on medication
* Recent hospitalisation (within the last 6 months)
* People with osteoarthritis.
* Anyone who has had a cardiovascular event in the last 30 years (angina, heart attack)
* People with a current clinical acute inflammatory condition.
* People who have practised sport with known vascular complications.
* Persons under guardianship or trusteeship
* Exclusion Criteria: withdraw of consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference of T cell metabolism between active and inactive participants | at day 0
  On the bloodwithdraw, level of T cells metabolism will be measured by using the SCENITH (Single Cell ENergetIc metabolism by profiling Translation inHibition) method
Difference of T cell metabolism between active and inactive participants | at day 0
  On the bloodwithdraw, level of T cells metabolism will be measured by RNA sequencing

SECONDARY OUTCOMES:
WHOQOLD-OLD Questionnaire | at day 0
  A low score reflects a poor quality of life, whereas a high score does not. 24 questions and 6 dimensions are assessed: physical state, psychological state, mobility, social life, environment and spirituality.
Capacity vitality | at day 0 and 14
  Evaluating all vitality capacity features regarding Bautmans 2022 guidelines
Neuromuscular parameters | at day 0 and 14
  Will be evaluated using HD-EMGs

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No